CLINICAL TRIAL: NCT03727425
Title: Robotic Bronchoscopy for Peripheral Pulmonary Lesions: A Multicenter Pilot and Feasibility Study
Brief Title: Robotic Bronchoscopy for Peripheral Pulmonary Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Auris Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-BR-0001
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Results first posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-10

CONDITIONS: Lung; Node
Keywords: Bronchoscopy; Robotic bronchoscopy; Lung cancer; Peripheral lesions
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Robotic assisted bronchoscopy (Experimental): Robotic assisted bronchoscopy procedures will be performed using the Monarch platform.
  Interventions: Device: Robotic assisted bronchoscopy

INTERVENTIONS:
Device: Robotic assisted bronchoscopy — Robotic assisted bronchoscopy of peripheral airways in human subjects for the purpose of biopsying peripheral lung lesions.
  Other Names: Monarch platform

SUMMARY:
In this study, the feasibility of performing robotic navigation of peripheral airways in human subjects for the purpose of biopsying peripheral lung lesions will be evaluated.

DETAILED DESCRIPTION:
Successful biopsy of peripheral pulmonary lesions remains a challenge due to a number of factors, one of which may be the ability to gain access to peripheral lesions due to the size and maneuverability of conventional bronchoscopes. In this study, the investigators will evaluate the feasibility of a new technique using a robotic endoscope with the Monarch navigational platform to both access and biopsy peripheral pulmonary lesions. The Monarch platform is a "robotic" assisted or electromechanical, software driven endoscopy system designed to be used by qualified physicians to provide bronchoscopic visualization of and access to patient airways for diagnostic and therapeutic procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Capable and willing to give informed consent
2. Acceptable candidate for an elective, non-emergent bronchoscopic procedure
3. Solid peripheral lung lesions suspected of malignancy, between 1-5cm in size identified on thin slice CT scan within 14 days of the intended bronchoscopy procedure
4. Lack bleeding disorders

Exclusion Criteria:

1. Medical contraindication to bronchoscopy
2. Patients with a subsolid nodule and/or ground-glass opacity lesions on pre-procedure chest CT
3. Patients with endobronchial involvement seen on chest CT
4. Lack fitness to undergo flexible bronchoscopy as determined by the bronchoscopist prior to procedure
5. Participation in any other investigational clinical trial (device or medication) 30 days before and throughout the duration of the study
6. Uncontrolled or irreversible coagulopathy
7. Female subjects who are pregnant or nursing or those of child-bearing potential refusing a pregnancy test
8. Have significant mediastinal lymphadenopathy on chest CT scan and/or PET CT abnormalities suggestive of advanced stage lung cancer with mediastinal lymph node involvement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, MD, Principal Investigator — Washington University School of Medicine; Gerard A Silvestri, MD, Principal Investigator — Medical University of South Carolina; Thomas R Gildea, MD, Principal Investigator — The Cleveland Clinic; Amit K Mahajan, MD, Principal Investigator — Innova Fairfax Hospital; Michael J Simoff, MD, Principal Investigator — Henry Ford Health System
Locations (5):
- United States (5):
  - Henry Ford Health System, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Innova Fairfax Hospital, Falls Church, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen AC, Pastis NJ Jr, Mahajan AK, Khandhar SJ, Simoff MJ, Machuzak MS, Cicenia J, Gildea TR, Silvestri GA. Robotic Bronchoscopy for Peripheral Pulmonary Lesions: A Multicenter Pilot and Feasibility Study (BENEFIT). Chest. 2021 Feb;159(2):845-852. doi: 10.1016/j.chest.2020.08.2047. Epub 2020 Aug 19. PMID 32822675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Robotic Assisted Bronchoscopy
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.1 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Not Hispanic or Latino | 42
  Ethnicity: Hispanic or Latino | 1
  Ethnicity: Not Reported | 11
  Ethnicity: Unknown | 1
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Device or Procedure Related Adverse Events
Description: Computed as the number of patients with device or procedure related adverse events divided by number of patients who underwent the robotic bronchoscopy procedure.
Time Frame: 24-84 hours post-procedure
Population: 54 patients underwent the robotic bronchoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 54
Participants | 2

2. Primary Outcome: Successful Navigation to Targeted Peripheral Pulmonary Lesions
Description: Successful navigation is confirmed using radial probe endobronchial ultrasound (R-EBUS). the R-EBUS will be inserted into the working channel of the endoscope and advanced beyond the tip of the inner scope as the inner scope is advanced into the lung periphery towards the targeted lesion. As the endoscope is guided towards the targeted lesion, R-EBUS will confirm successful lesion localization prior to biopsies being performed.
Time Frame: During the procedure, approximately 1 hour
Population: Radial probe endobronchial ultrasound was available in 53/54 cases.
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 53
Participants | 51

3. Secondary Outcome: Incidence of Complications Unrelated to Device
Description: Computed as the number of patients with events unrelated to device or procedure divided by number of patients who underwent the robotic bronchoscopy procedure.
Time Frame: 24-84 hours post-procedure
Population: 54 patients underwent the robotic bronchoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 54
Participants | 0

4. Secondary Outcome: Time to R-EBUS Confirmation (Lesion Localization)
Description: Defined by the time the robotic bronchoscope is inserted into the oropharynx until the localization of the targeted lesion is confirmed by REBUS.
Time Frame: During the procedure, approximately 1 hour
Population: Radial probe endobronchial ultrasound was available in 53/54 cases.
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 53
Minutes | 13 [25 to 75]

5. Secondary Outcome: Total Procedure Time
Description: Defined by the time the robotic bronchoscope is inserted into the oropharynx until the time a biopsy tool is removed.
Time Frame: During the procedure
Population: 54 patients underwent the robotic bronchoscopy procedure
Measure: Mean (Inter-Quartile Range); unit: Minutes
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 54
Minutes | 51 [25 to 75]

6. Secondary Outcome: Diagnostic Yield
Description: Determined from the results of the bronchoscopy.
Time Frame: Data was collected (as part of standard of care) through 1-year for calculation of diagnostic yield.
Population: 54 patients underwent the robotic bronchoscopy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Robotic Assisted Bronchoscopy
Number analyzed (Participants) | 54
Participants | 40

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from time of procedure through 84 hours post procedure.
Arm/Group | Robotic Assisted Bronchoscopy
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 2/55
Other Adverse Events (participants affected / at risk) | 0/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Robotic Assisted Bronchoscopy (N=55)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT03727425/Prot_SAP_001.pdf